CLINICAL TRIAL: NCT04161547
Title: A Phase I, Ascending Multiple-dose Clinical Trial of CSPCHA115 Capsules to Evaluate the Tolerability and Pharmacokinetics in Chinese Healthy Volunteers
Brief Title: Tolerability and Pharmacokinetics of CSPCHA115 Capsules in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HA116201903/PRO I-MAD
Record Dates: First submitted 2019-10-29; First posted 2019-11-13 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: CSPCHA115; Asthma; CRTH2
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A1: CSPCHA115 100 mg (Experimental): CSPCHA115 100 mg or placebo administered orally in the fasted state for 7 days.
  * Eight subjects will receive CSPCHA115
  * Two subjects will receive matching placebo
  Interventions: Drug: CSPCHA115 100 mg; Matching placebo 100 mg
- Cohort A2: CSPCHA115 200 mg (Experimental): CSPCHA115 200 mg or placebo administered orally in the fasted state for 7 days.
  * Eight subjects will receive CSPCHA115
  * Two subjects will receive matching placebo
  Interventions: Drug: CSPCHA115 200 mg; Matching placebo 200 mg
- Cohort A3: CSPCHA115 400 mg (Experimental): CSPCHA115 400 mg or placebo administered orally in the fasted state for 7 days.
  * Eight subjects will receive CSPCHA115
  * Two subjects will receive matching placebo
  Interventions: Drug: CSPCHA115 400 mg; Matching placebo 400 mg
- Cohort A4: CSPCHA115 600 mg (Experimental): CSPCHA115 600 mg or placebo administered orally in the fasted state for 7 days.
  * Eight subjects will receive CSPCHA115
  * Two subjects will receive matching placebo
  Interventions: Drug: CSPCHA115 600 mg; Matching placebo 600 mg

INTERVENTIONS:
Drug: CSPCHA115 100 mg; Matching placebo 100 mg — CSPCHA115 100 mg once daily in the fasted state for 7 days; Matching placebo 100 mg once daily in the fasted state for 7 days.
  Arms: Cohort A1: CSPCHA115 100 mg
Drug: CSPCHA115 200 mg; Matching placebo 200 mg — CSPCHA115 200 mg once daily in the fasted state for 7 days; Matching placebo 200 mg once daily in the fasted state for 7 days.
  Arms: Cohort A2: CSPCHA115 200 mg
Drug: CSPCHA115 400 mg; Matching placebo 400 mg — CSPCHA115 400 mg once daily in the fasted state for 7 days; Matching placebo 400 mg once daily in the fasted state for 7 days.
  Arms: Cohort A3: CSPCHA115 400 mg
Drug: CSPCHA115 600 mg; Matching placebo 600 mg — CSPCHA115 600 mg once daily in the fasted state for 7 days; Matching placebo 600 mg once daily in the fasted state for 7 days.
  Arms: Cohort A4: CSPCHA115 600 mg

SUMMARY:
A randomized, single-center, double-blind, ascending multiple-dose, placebo-controlled study to evaluate the tolerability and pharmacokinetics of CSPCHA115 capsules in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 45 years old, male or female;
* Bodyweight≥45.0 kg (female) or 50.0 kg (male), 19 kg/m^2 ≤ Body Mass Index（BMI ）≤ 26 kg/m^2;
* The female subjects are not during pregnancy or lactation; the male subjects have no sperm donation plan from the signing of the informed consent form to 1 month after the completion of the study. The subjects and their partners agree to use effective non-hormonal contraceptives (such as condoms, drug-free IUDs, etc.) from the day signing the informed consent form to 1 month after the completion of the study, or had taken permanent contraceptives (such as bilateral tubal ligation, vasectomy, etc.);
* Subjects voluntarily sign the informed consent form, and are able to complete the trial according to the protocol;

Exclusion Criteria:

Those who conform to one of the following provisions shall not be included in the group;

* A clear history of neurological or mental disorders (including seizures, dementia, depression or biphasic affective disorders, etc.); immunodeficient or immunosuppressive diseases, malignant tumor diseases; cardiovascular, liver and kidney, endocrine, respiratory, blood, digestive system and other chronic diseases;
* Subjects who underwent large surgical operations within 6 months before signing the informed consent (such as coronary artery bypass grafting, hepatorenectomy, nephrectomy, gynecological surgery, etc.), and those with acute neurological, digestive, respiratory, circulation, endocrine, blood and other systemic diseases within 3 months before signing the informed consent form may affect the absorption, distribution, metabolism and excretion of drugs;
* Subjects with allergic constitutions, or who are allergic to more than 1 drug, or had other known serious allergic reactions;
* Subjects who did not meet the health criteria during the screening period, including abnormal vital signs; QTc interval ≥ 450 ms (male) or 470ms (female), prolongation of QTc interval, or other abnormal clinical significance of electrocardiogram (ECG); the results of physical examination, laboratory examination and so on are abnormal and have clinical significance.
* One of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), human immunodeficiency virus antibody (Anti-HIV) and Treponema pallidum antibody (Anti-TP) was positive;
* Any prescription drugs, non-prescription drugs, biological products, the Chinese patent medicines, herbs, vitamin dietary supplements, and health-care products (other than external use), oral long-acting contraceptives or embedded long-acting contraceptives were used regularly within 2 weeks before the signing of the informed consent form;
* A history of alcoholism, or alcohol test positive at screening;
* The average daily smoking volume was more than 5 within 6 months before signing the informed consent form;
* Drug abuse within 1 year before signing the informed consent form, or urine test positive for drugs at screening;
* Subjects who were accustomed to excessive caffeine drinks or foods that may affect drug metabolism within 4 weeks prior to the signing of the informed consent form;
* Subjects who lost blood or donated more than 200 ml within 8 weeks before signing the informed consent form, or who planned to donate blood within 1 month after the completion of the study;
* Subjects who plan to undergo surgery during the trial period, or those who plan to take part in strenuous exercise during the trial period;
* Subjects who are participating in other clinical trials, or who have participated in clinical trial about any other drugs or devices within 3 months before signing the informed consent form;
* Not suitable for this clinical trial judged by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Number and incidence of subjects with Adverse Events (AEs) | 12 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Number of subjects with clinically significant symptoms abnormalities | 10 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Number of subjects with clinically significant vital sign abnormalities | 10 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Number of subjects with clinically significant physical examination abnormalities | 10 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Number of subjects with clinically significant laboratory abnormalities | 10 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Number of subjects with clinically significant electrocardiograms (ECGs) abnormalities | 10 days after drug administration
  To evaluate the safety and tolerability after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Time to reach maximum observed concentration (Tmax) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Maximum observed concentration (Cmax) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Area under the concentration-time curve from time 0 to 24h (AUC0-24h) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Tmax at steady state (Tss max) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Cmax at steady state (Css max) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Cmin at steady state (Css min) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Average concentration at steady state (Css av) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
AUC at steady state (AUCss) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Elimination half-life (t1/2) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Apparent clearance at steady state (CLss/F) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Apparent volume of distribution (Vz/F) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Fluctuation coefficient (DF) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg
Accumulation ratio (Rac) | Day 1(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours); Day 5(Pre-dose); Day 6(Pre-dose); Day 7(Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours) after drug administration
  To evaluate the pharmacokinetics after repeated administrations of CSPCHA115 capsules 100, 200, 400 and 600 mg

CONTACTS AND LOCATIONS:
Overall Officials: Xuefang Xia, Study Director — Department of Medicine, CSPC Clinical Development Division
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China